CLINICAL TRIAL: NCT02157688
Title: Role of Staphylococcus Aureus on Folliculitis Decalvans. A Comparative Bacteriological Study.
Brief Title: Impact of Staphylococcus Aureus on Folliculitis Decalvans
Acronym: SAFE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: SAFE Folliculitis Decalvans
Record Dates: First submitted 2014-05-14; First posted 2014-06-06 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2015-03

CONDITIONS: Folliculitis Decalvans; Staphylococcus Aureus
Keywords: folliculitis decalvans; Staphylococcus Aureus; antibiotics
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case: Patient with a folliculitis Decalvans
  Interventions: Other: no intervention : case control study
- control: Control without folliculitis decalvans
  Interventions: Other: no intervention : case control study

INTERVENTIONS:
Other: no intervention : case control study

SUMMARY:
The folliculitis decalvans (FD) is an orphan disease , common in consultation specialized on scalp. This disease is currently not curable, responsible for significant for patients. The pathophysiology is poorly understood, Staphylococcus aureus (SA) appears to play a role, never previously studied, and the study will attempt to clarify it.

Controversies in the literature on the pathophysiological hypotheses can be summed up as follows :

FD is it an infectious folliculitis where SA (almost always found on the lesions plays a direct role possibly aided by a lack of local immune protection , or is it a pustular inflammatory unknown cause where the SA has no direct role but is a cofactor or a simple germ superinfection.

Our study has plans to bring new evidence to help decide between these two opposite but not mutually exclusive concepts .

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 yo)
* Alopecia
* folliculitis decalvans
* At least 6 months of evolution
* no antibiotics
* presence of pustules and crusts
* Adult (>18 yo)

Exclusion Criteria:

* immunosuppression
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with Folliculitis Decalvans
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
presence of Staphylococcus Aureus in cutaneous biopsies (at least one colony) | 1 day
  The primary endpoint is the presence of Staphylococcus Aureus in cutaneous biopsies before any therapy and notably antibiotics.

SECONDARY OUTCOMES:
presence of Staphylococcus Aureus in cutaneous biopsies (at least one colony) after treatment | 10 weeks
presence of Staphylococcus Aureus in nasal swab (at least one colony) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, Paris, France

REFERENCES:
- [Derived] Matard B, Donay JL, Resche-Rigon M, Tristan A, Farhi D, Rousseau C, Mercier-Delarue S, Cavelier-Balloy B, Assouly P, Petit A, Bagot M, Reygagne P. Folliculitis decalvans is characterized by a persistent, abnormal subepidermal microbiota. Exp Dermatol. 2020 Mar;29(3):295-298. doi: 10.1111/exd.13916. Epub 2019 May 15. PMID 30907453